CLINICAL TRIAL: NCT04110197
Title: Demographic Outcomes, and Health Care Resources in Newly Diagnosed Non Valvular AF Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Taha Mohamed, resident doctor, Assiut University
Other Study IDs: non valvular AF
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Non Valvular AF ,AF

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To describe the patterns of care of newly diagnosed patients with NVAF vs VAF in the first-line, second-line and beyond second line setting, including, treatment plan, regimen, dosing, duration of treatment, and reason for interruption and termination along with treatment switching at any point of treatment, regardless if the patients are considered of first line, second line or further within the treatments.
2. To describe the clinical outcomes (stroke/systemic embolism, bleeding complications, as well as cause-specific and all-cause mortality) with NVAF vs VAF.
3. To describe the values and distribution of International normalized ratio (INR) in patients who received VKAs and to assess the influence of Time in therapeutic range (TTR) and INR history on clinical outcomes (stroke/systemic embolism, bleeding complications) with NVAF vs VAF.
4. To evaluate AF-related healthcare resource utilization and direct costs associated with the management of AF patients with NVAF vs VAF.

and To describe the baseline clinical and demographic characteristics as well as risk factors among patients newly diagnosed with NVAF versus VAF.

ELIGIBILITY:
Inclusion Criteria:

* 1. All male or female patients aged 18 years and older at the date of inclusion.

  2. Patient newly diagnosed [within the recruitment period (estimated to be 6 months) and 90 days before the baseline visit] with atrial fibrillation (AF) and for whom treatment has started by the caring physician for the prevention of stroke/systemic embolism.

  3. Signed informed consent.

Exclusion Criteria:

* 2. Severe psychiatric illness or other disease or circumstances that could compromise participation in the study. Patients will not be enrolled if major difficulties with follow-up will be anticipated, for example, patients with no valid residency permit or those planning to leave the country before the next scheduled follow-up.

  3. Current participation in an interventional clinical trial at baseline. 4. AF with a generally reversible cause defined as non-cardiac surgery, post-cardiac surgery (AF within 3 months after surgery), hyperthyroidism, pulmonary embolism, pneumonia and acute myocardial infarction.

  5. Mechanical heart valves or valve disease expected to require valve replacement.

  6. A medical condition other than AF for which chronic use of VKA/NOAC is indicated.

  7. Pregnant or breast-feeding women. Pregnancy to be ruled out according normal practice method of each site.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study to be carried out in Assiut University Heart Hospital.
  The study is designed to capture real-world evidence (RWE) on patients' characteristics and the clinical management of patients with with NVAF vs VAF. All consecutive patients that are newly diagnosed with NVAF within the recruitment period (estimated to be 6 months) and 90 days before baseline visit and who meet the study inclusion/exclusion criteria will be invited to participate in the study. The study periods may be revised based on recruitment rate.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
● Stroke: hemorrhagic or ischemic; ● Transient Ischemic Attack (TIA); ● Systemic embolism; ● Bleeding events (see definitions and categories below); ● Myocardial infarction; ● All-cause mortality. | 6 monthes
  * Acute clinically overt bleeding accompanied by one or more of the following:
  * A decrease in hemoglobin (Hgb) of 2 g/dL or more over a 24-hour period;
  * A transfusion of 2 or more units of packed red blood cells.
  * Bleeding that occurs in at least one of the following critical sites:
  * Intracranial;
  * Intra-spinal;
  * Intraocular (within the corpus of the eye; thus, a conjunctival bleed is not an intraocular bleed);
  * Pericardial;
  * Intra-articular;
  * Intramuscular with compartment syndrome;
  * Retroperitoneal.
  * Bleeding that is fatal.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
demographic base line , medical history clinical picture and complications treatment compliance follow up hospital admission and health resources
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: demographic base line , medical history clinical picture and complications treatment compliance follow up hospital admission and health resources